CLINICAL TRIAL: NCT02292758
Title: BOND-3: A Randomized, Double-Blind, Placebo-Controlled Phase II Trial of Irinotecan, Cetuximab, and Bevacizumab Compared With Irinotecan, Cetuximab, and Placebo in RAS-Wildtype, Irinotecan-Refractory, Metastatic Colorectal Cancer
Brief Title: Irinotecan and Cetuximab With or Without Bevacizumab in Treating Patients With RAS Wild-Type Locally Advanced or Metastatic Colorectal Cancer That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Academic and Community Cancer Research United (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RU021302I; NCI-2016-02063 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RU021302I (Other: Academic and Community Cancer Research United); P30CA015083 (NIH)
Record Dates: First submitted 2014-11-13; First posted 2014-11-17 (Estimated); Results first posted 2020-02-28 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2019-08

CONDITIONS: Colorectal Adenocarcinoma; RAS Wild Type; Stage IV Colorectal Cancer AJCC v7; Stage IVA Colorectal Cancer AJCC v7; Stage IVB Colorectal Cancer AJCC v7
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Cetuximab; Irinotecan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (cetuximab, bevacizumab, irinotecan) (Experimental): Patients receive cetuximab IV over 90-120 minutes, bevacizumab IV over 30-90 minutes, and irinotecan IV over 90 minutes on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Biological: Cetuximab; Drug: Irinotecan; Other: Laboratory Biomarker Analysis
- Arm II (cetuximab, placebo, irinotecan) (Active Comparator): Patients receive cetuximab IV over 90-120 minutes, placebo IV over 30-90 minutes, and irinotecan IV over 90 minutes on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Cetuximab; Drug: Irinotecan; Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501
  Arms: Arm I (cetuximab, bevacizumab, irinotecan)
Biological: Cetuximab — Given IV
  Other Names: Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
Drug: Irinotecan — Given IV
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given IV
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (cetuximab, placebo, irinotecan)

SUMMARY:
This randomized phase II trial studies how well irinotecan and cetuximab with or without bevacizumab work in treating patients with RAS wild-type colorectal cancer that has spread to other places in the body (locally advanced/metastatic) and cannot be removed by surgery. Irinotecan may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Immunotherapy with monoclonal antibodies, such as cetuximab and bevacizumab, may help the body?s immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving irinotecan and cetuximab with or without bevacizumab may work betting in treating patients with colorectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess and compare the progression-free survival (PFS) of patients receiving irinotecan, cetuximab, and bevacizumab with patients receiving irinotecan, cetuximab and placebo, in the population of patients with RAS wild-type, irinotecan-refractory metastatic colorectal cancer (mCRC) who also previously received bevacizumab in at least one prior line therapy.

SECONDARY OBJECTIVES:

I. To assess the adverse event (AE) profile and safety of the proposed treatment in this population.

II. To assess and compare the overall survival (OS) between treatment arms in this population.

III. To assess and compare the disease control rate (DCR) between treatment arms in this population.

IV. To assess and compare the overall response rate (ORR) between treatment arms in this population.

V. To assess and compare the duration of response between treatment arms in this population.

VI. To assess and compare time to treatment failure between treatment arms in this population.

VII. To assess relative dose intensity of treatment agents between treatment arms in this population.

CORRELATIVE OBJECTIVES:

I. Determine the change in genotype concentrations of prespecified gene mutations in circulating cell-free deoxyribonucleic acid (DNA) (cfDNA) collected serially during protocol treatment.

II. Explore the predictive value of pretreatment mutation status, germline single nucleotide polymorphisms (SNPs), and gene expression signatures for cetuximab sensitivity and resistance.

III. Explore the predictive value of dynamic changes in mutation status and gene expression signatures for cetuximab sensitivity and resistance.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive cetuximab intravenously (IV) over 90-120 minutes, bevacizumab IV over 30-90 minutes, and irinotecan IV over 90 minutes on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive cetuximab IV over 90-120 minutes, placebo IV over 30-90 minutes, and irinotecan IV over 90 minutes on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or locally advanced (unresectable) colorectal cancer with histological confirmation of adenocarcinoma
* Measurable disease
* RAS wild-type tumor; Note: evidence of EGFR expression in the tumor is not required
* Previous failure of at least one fluoropyrimidine- and irinotecan-containing chemotherapy regimen for metastatic disease; Note: previous failure is defined as disease progression while receiving treatment or within 6 weeks after the last dose of irinotecan; failure for this assessment is defined as any enlargement of measurable or assessable lesion(s) or the development of any new lesion; a rising tumor marker alone is not sufficient to define failure; patients can have received irinotecan in any previous line of therapy
* Treatment with bevacizumab in at least one prior line of therapy for metastatic disease
* Negative serum or urine pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Eastern Cooperative Oncology Group (ECOG) performance status (PS): 0 or 1
* Total serum bilirubin =< institutional upper limit of normal (ULN) obtained =<14 days prior to randomization
* Absolute neutrophil count (ANC) >= 1500/mm^3 obtained =<14 days prior to randomization
* Platelet count >= 100,000/mm^3 obtained =<14 days prior to randomization
* Hemoglobin >= 9.0 g/dL (hemoglobin may be supported by transfusion) obtained =<14 days prior to randomization
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 2.5 x ULN (=< 5 x ULN for subjects with liver involvement of their cancer) obtained =<14 days prior to randomization
* Creatinine within institutional limits of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal obtained =<14 days prior to randomization
* Urinary protein =< 1+ obtained =<14 days prior to randomization

  * Patients discovered to have >= 2+ proteinuria must have a spot urine protein:creatinine ratio (UPCR) < 1.0
* Partial thromboplastin time (PTT) =< 1 x institutional ULN and international normalized ratio (INR) =< 1.5 , unless participant is on full dose anticoagulation therapy obtained =<14 days prior to randomization; patients on full-dose anticoagulation are eligible if the following criteria are met:

  * Patient has an in-range INR (usually 2-3) on a stable dose of warfarin or other anticoagulant =< 14 days or is on a stable dose of low molecular weight heparin
  * Patient has no active bleeding or pathological condition that carries a high risk of bleeding (i.e., tumor involving major vessels or known varices)
  * Patients receiving anti-platelet agents are eligible; in addition, patients who are on daily prophylactic aspirin or anticoagulation for atrial fibrillation are eligible
* Life expectancy > 3 months
* Provide informed written consent
* Willing to provide blood samples for mandatory correlative and research purposes
* Willing to provide tissue and blood samples for mandatory banking purposes
* Any major surgery or open biopsy completed >= 4 weeks prior to randomization
* Any minor surgery or core biopsy completed >= 1 week prior to randomization and patient must have fully recovered from the procedure; Note: insertion of a vascular access device is not considered major or minor surgery

Exclusion Criteria:

* Presence of a RAS mutation in exons 2, 3, or 4 of KRAS or NRAS (patients with mutations in exons 2, 3, or 4 of KRAS and/or NRAS are excluded)
* Prior treatment with cetuximab or panitumumab
* Prior intolerance to irinotecan and/or bevacizumab despite dose reduction
* Known or suspected brain or central nervous system (CNS) metastases, or carcinomatous meningitis
* Active, uncontrolled infection, including hepatitis B, hepatitis C
* Concurrent anti-cancer therapy, including chemotherapy agents, targeted agents, or biological agents not otherwise specified in this protocol
* Anti-cancer therapy =< 14 days prior to randomization
* Prior radiotherapy to > 25% of bone marrow; Note: standard rectal cancer chemoradiation will not exclude subject from study protocol
* Radiation therapy =< 2 weeks prior to randomization
* Any of the following:

  * Pregnant women
  * Nursing women
  * Men or women of childbearing potential who are unwilling to employ adequate contraception
* Co-morbid systemic illnesses or other severe concurrent disease, history of any psychiatric or addictive disorder, or laboratory abnormality, which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Patients known to be human immunodeficiency virus (HIV) positive
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, symptomatic pulmonary fibrosis or interstitial pneumonitis, or psychiatric illness/social situations that, in the opinion of the investigator, may increase the risks associated with study participation or study treatment, or may interfere with the conduct of the study or the interpretation of the study results
* Receiving any other investigational agent which would be considered as a treatment for the primary neoplasm
* Other active malignancy =< 3 years prior to registration; EXCEPTIONS: non-melanoma skin cancer, prostatic intraepithelial neoplasia without evidence of prostate cancer, lobular carcinoma in situ in one breast, or carcinoma-in-situ of the cervix that has been treated
* History of prior malignancy for which patient is receiving other specific treatment for their cancer
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to irinotecan, cetuximab, and/or bevacizumab that led to discontinuation of those agents
* Significant history of bleeding events or pre-existing bleeding diathesis =< 6 months of randomization (unless the source of bleeding has been resected)
* History of gastrointestinal perforation =< 12 months prior to randomization
* Predisposing colonic or small bowel disorders in which the symptoms are uncontrolled as indicated by baseline pattern of > 3 loose stools daily in subjects without a colostomy or ileostomy; subjects with a colostomy or ileostomy may be entered at investigator discretion
* Arterial thrombotic events =< 6 months prior to randomization; Note: this includes transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina or angina requiring surgical or medical intervention in the past 6 months, or myocardial infarction (MI)
* Clinically significant peripheral artery disease (e.g., claudication with < 1 block) or any other arterial thrombotic event
* Serious or non-healing wound, ulcer, or bone fracture
* History of hypertension not well-controlled (>= 160/90) even though on a regimen of anti-hypertensive therapy
* Evidence of Gilbert?s syndrome or known homozygosity for the UGT1A1*28 allele (special screening not required)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2019-03-20 (Actual); Study Completion 2019-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimmie Ng, Principal Investigator — Academic and Community Cancer Research United
Locations (13):
- United States (13):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Cancer Center of Kansas - Wichita, Wichita, Kansas
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Michigan Cancer Research Consortium NCORP, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Heartland Regional Medical Center, Saint Joseph, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - New Hampshire Oncology Hematology PA-Hooksett, Hooksett, New Hampshire
  - State University of New York Upstate Medical University, Syracuse, New York
  - Saint Vincent Regional Cancer Center CCOP, Green Bay, Wisconsin

REFERENCES:
- [Derived] Lipsyc-Sharf M, Ou FS, Yurgelun MB, Rubinson DA, Schrag D, Dakhil SR, Stella PJ, Weckstein DJ, Wender DB, Faggen M, Zemla TJ, Heying EN, Schuetz SR, Noble S, Meyerhardt JA, Bekaii-Saab T, Fuchs CS, Ng K. Cetuximab and Irinotecan With or Without Bevacizumab in Refractory Metastatic Colorectal Cancer: BOND-3, an ACCRU Network Randomized Clinical Trial. Oncologist. 2022 Apr 5;27(4):292-298. doi: 10.1093/oncolo/oyab025. PMID 35380713

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Irinotecan, Cetuximab, Bevacizumab): Patients receive 500 mg/m^2 cetuximab IV over 90-120 minutes, 5 mg/kg bevacizumab IV over 30-90 minutes, and 180 mg/m^2 irinotecan IV over 90 minutes on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.
- Arm II (Irinotecan, Cetuximab, Placebo): Patients receive 500 mg/m^2 cetuximab IV over 90-120 minutes, 5 mg/kg placebo IV over 30-90 minutes, and 180 mg/m^2 irinotecan IV over 90 minutes on day 1. Cycles repeat every 14 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm I (Irinotecan, Cetuximab, Bevacizumab) | Arm II (Irinotecan, Cetuximab, Placebo)
Started | 19 | 17
Completed | 19 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Irinotecan, Cetuximab, Bevacizumab) | Arm II (Irinotecan, Cetuximab, Placebo) | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Median (Full Range); unit: years] | 58 [41 to 71] | 54 [39 to 82] | 55 [39 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 10 | 10 | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 15 | 15 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group PS Scale: 0)Fully active, able to carry on all pre-disease performance without restriction; 1)Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2)Ambulatory and capable of all selfcare but unable to carry out any work activities. Up and about more than 50% of waking hours; 3)Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours; 4)Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  Participants
    0 | 14 | 12 | 26
    1 | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: The distribution of PFS by group will be estimated using the method of Kaplan-Meier. Median by treatment group with confidence intervals will be estimated based on Kaplan-Meier curves. The hazard ratio (HR) with confidence interval will be estimated based on stratified Cox models (stratified by levels of stratification factors), without and with adjusting for baseline clinical/pathological factors. Progression (PD) is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. PD: Any new lesion or increase by ≥50% of previously involved sites from nadir).
Time Frame: From the date of randomization to the date of 1st documented disease progression or death due to any cause, whichever occurs first, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Irinotecan, Cetuximab, Bevacizumab) | Arm II (Irinotecan, Cetuximab, Placebo)
Number analyzed (Participants) | 19 | 17
months | 9.7 [7.1 to 13.7] | 5.5 [3.8 to 10.2]
Statistical Analysis 1: Comparison: Arm I (Irinotecan, Cetuximab, Bevacizumab) vs Arm II (Irinotecan, Cetuximab, Placebo); Test type: Superiority; p = 0.7609, Log Rank; Hazard Ratio (HR) = 0.912, 95% CI 2-sided [0.431 to 1.930] — Unadjusted HR; Model stratified by: prior bevacizumab (Y vs N) and prior lines of chemotherapy (1 vs 2+)
Statistical Analysis 2: Comparison: Arm I (Irinotecan, Cetuximab, Bevacizumab) vs Arm II (Irinotecan, Cetuximab, Placebo); Test type: Superiority; Hazard Ratio (HR) = 0.642, 95% CI 2-sided [0.249 to 1.656] — Adjusted HR; Model adjusted by: age, gender, race (white vs others), number of metastatic sites (1 vs 2 vs 3+), ECOG PS (0 vs 1), tumor site (colon, rectum/rectosigmoid, multiple)

2. Primary Outcome: 6-month and 12-month Progression-free Survival (PFS) Rates
Description: The distribution of PFS by group will be estimated using the method of Kaplan-Meier. Six and 12 month PFS rates by treatment group with confidence intervals will be estimated based on Kaplan-Meier curves. The hazard ratio (HR) with confidence interval will be estimated based on stratified Cox models (stratified by levels of stratification factors), without and with adjusting for baseline clinical/pathological factors. Progression (PD) is defined according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. PD: Any new lesion or increase by ≥50% of previously involved sites from nadir).
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Irinotecan, Cetuximab, Bevacizumab) | Arm II (Irinotecan, Cetuximab, Placebo)
Number analyzed (Participants) | 19 | 17
percentage of participants
  6-month PFS rate | 76.5 [58.7 to 99.5] | 41.2 [23.3 to 72.7]
  12-month PFS rate | 27.5 [12.3 to 61.2] | 17.6 [6.3 to 49.3]

3. Secondary Outcome: Number of Participants Who Experienced at Least One Grade 3 or Higher Adverse Events
Description: The number of participants who experienced at least one grade 3 or higher adverse events assessed by National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 30 days from last dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Irinotecan, Cetuximab, Bevacizumab) | Arm II (Irinotecan, Cetuximab, Placebo)
Number analyzed (Participants) | 19 | 17
Participants | 9 | 6

4. Secondary Outcome: Overall Survival (OS)
Description: The distribution of OS by group will be estimated using the method of Kaplan-Meier. Median OS by treatment group with confidence intervals will be estimated based on Kaplan-Meier curves. The HR with confidence interval will be estimated based on stratified Cox models (stratified by levels of stratification factors), without and with adjusting for baseline clinical/pathological factors.
Time Frame: From randomization to the date of death due to any cause, assessed up to 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Irinotecan, Cetuximab, Bevacizumab) | Arm II (Irinotecan, Cetuximab, Placebo)
Number analyzed (Participants) | 19 | 17
months | 19.7 [14.9 to NA] — The 95% confidence interval upper limit was not reached (i.e. under the level of detection). | 10.2 [7.9 to 16.0]
Statistical Analysis 1: Comparison: Arm I (Irinotecan, Cetuximab, Bevacizumab) vs Arm II (Irinotecan, Cetuximab, Placebo); Test type: Superiority; p = 0.0446, Log Rank; Hazard Ratio (HR) = 0.471, 95% CI 2-sided [0.209 to 1.062] — Unadjusted HR; Model stratified by: prior bevacizumab (Y vs N) and prior lines of chemotherapy (1 vs 2+)
Statistical Analysis 2: Comparison: Arm I (Irinotecan, Cetuximab, Bevacizumab) vs Arm II (Irinotecan, Cetuximab, Placebo); Test type: Superiority; Hazard Ratio (HR) = 0.406, 95% CI 2-sided [0.151 to 1.089] — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: 12-month, 18-month, and 24-month Overall Survival (OS) Rates
Description: The distribution of OS by group will be estimated using the method of Kaplan-Meier. Twelve, 18- and 24-month survival rates by treatment group with confidence intervals will be estimated based on Kaplan-Meier curves. The HR with confidence interval will be estimated based on stratified Cox models (stratified by levels of stratification factors), without and with adjusting for baseline clinical/pathological factors.
Time Frame: From randomization to the date of death due to any cause, assessed up to 24 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Irinotecan, Cetuximab, Bevacizumab) | Arm II (Irinotecan, Cetuximab, Placebo)
Number analyzed (Participants) | 19 | 17
percentage of participants
  12-month OS rate | 77.2 [59.7 to 99.8] | 47.1 [28.4 to 77.9]
  18-month OS rate | 56.1 [36.0 to 87.5] | 11.8 [3.2 to 43.2]
  24-month OS rate | 14.0 [2.4 to 81.1] | 5.9 [0.9 to 39.4]

6. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control is defined as maintaining Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) as the tumor assessment result during the defined time window. DCR (percentage) is defined as number of patients with success of disease control divided by total number of patients in the analysis population multiplied by 100, excluding patients who refuse treatment before the initiation of any treatment. CR: Disappearance of all evidence of disease, PR: Regression of measurable disease and no new sites, PD: Any new lesion or increase by ≥50% of previously involved sites from nadir, SD: Neither sufficient shrinkage to qualify for PR, nor sufficient increase to qualify for PD taking as reference the MSD
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Irinotecan, Cetuximab, Bevacizumab) | Arm II (Irinotecan, Cetuximab, Placebo)
Number analyzed (Participants) | 19 | 17
percentage of participants | 68.4 | 52.9
Statistical Analysis 1: Comparison: Arm I (Irinotecan, Cetuximab, Bevacizumab) vs Arm II (Irinotecan, Cetuximab, Placebo); Test type: Superiority; p = 0.3415, Chi-squared

7. Secondary Outcome: Overall Response Rate (ORR)
Description: The response rate (percentage) is the percent of participants whose best response was Complete Response (CR) or Partial Response (PR) as defined by RECIST 1.1 criteria. Percentage of successes will be estimated by 100 times the number of successes divided by the total number of evaluable patients. Response rates (including complete and partial response) will be tested using Fisher's exact test. CR: Disappearance of all evidence of disease, PR: Regression of measurable disease and no new sites
Time Frame: Up to 2 years
Measure: Number; unit: percentage of participants
Arm/Group | Arm I (Irinotecan, Cetuximab, Bevacizumab) | Arm II (Irinotecan, Cetuximab, Placebo)
Number analyzed (Participants) | 19 | 17
percentage of participants | 36.8 | 11.8
Statistical Analysis 1: Comparison: Arm I (Irinotecan, Cetuximab, Bevacizumab) vs Arm II (Irinotecan, Cetuximab, Placebo); Test type: Superiority; p = 0.1279, Fisher Exact

8. Secondary Outcome: Duration of Response (DOR)
Description: The distribution of DOR by treatment group will be estimated using the method of Kaplan-Meier. Six and 12 month durable response (i.e. maintaining CR or PR without progressive disease [PD]) rates by treatment group with confidence intervals will be estimated based on Kaplan-Meier curves. The HR with confidence interval will be estimated based on stratified Cox models (stratified by levels of stratification factors), without and with adjusting for baseline clinical/pathological factors.CR: Disappearance of all evidence of disease, PR: Regression of measurable disease and no new sites, PD: Any new lesion or increase by ≥50% of previously involved sites from nadir
Time Frame: From the date of first tumor assessment with the response status being CR or PR to the date of 1st documented progressive disease, assessed up to 12 months
Population: Participants who responded to treatment (CR or PR) are included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Irinotecan, Cetuximab, Bevacizumab) | Arm II (Irinotecan, Cetuximab, Placebo)
Number analyzed (Participants) | 7 | 2
months | 9.2 [3.5 to 14.8] | 9.7 [3.7 to 15.6]
Statistical Analysis 1: Comparison: Arm I (Irinotecan, Cetuximab, Bevacizumab) vs Arm II (Irinotecan, Cetuximab, Placebo); Test type: Superiority; p = 0.447, Log Rank

9. Secondary Outcome: Percentage of Participants With Treatment Failure at 6 Months
Description: TTF is defined as the time from the date of randomization to the date of treatment discontinuation due to PD, death, or severe AE. The distribution of TTF by treatment group will be estimated using the method of Kaplan-Meier. Six month event-free rates by treatment group with confidence intervals will be estimated based on Kaplan-Meier curves. The HR with confidence interval will be estimated based on stratified Cox models (stratified by levels of stratification factors), without and with adjusting for baseline clinical/pathological factors. PD: Any new lesion or increase by ≥50% of previously involved sites from nadir
Time Frame: assessed at 6 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Irinotecan, Cetuximab, Bevacizumab) | Arm II (Irinotecan, Cetuximab, Placebo)
Number analyzed (Participants) | 19 | 17
percentage of participants | 72.7 [54.9 to 96.3] | 38.4 [19.7 to 74.8]
Statistical Analysis 1: Comparison: Arm I (Irinotecan, Cetuximab, Bevacizumab) vs Arm II (Irinotecan, Cetuximab, Placebo); Test type: Superiority; p = 0.3738, Log Rank; Hazard Ratio (HR) = 0.755, 95% CI 2-sided [0.345 to 1.655] — Unadjusted HR; Model stratified by: prior bevacizumab (Y vs N) and prior lines of chemotherapy (1 vs 2+)

10. Secondary Outcome: Relative Dose Intensity (RDI)
Description: RDI is defined as the total dose of protocol therapy a patient actually received (i.e., summation of actually received dose at each cycle) divided by the total planned dose (i.e., summation of planned dose level at each cycle) multiplied by 100. Separate RDIs will be calculated for irinotecan and cetuximab. Agent-specific RDI will be summarized by medians, and min and max values, all of which will be compared between the two treatment groups by the Wilcoxon Rank sum test.
Time Frame: Up to 2 years
Measure: Median (Full Range); unit: percentage of dose received
Arm/Group | Arm I (Irinotecan, Cetuximab, Bevacizumab) | Arm II (Irinotecan, Cetuximab, Placebo)
Number analyzed (Participants) | 19 | 17
percentage of dose received
  Cetuximab | 98.5 [60.9 to 152.9] | 95.5 [40.0 to 103.4]
  Irinotecan | 89 [40.8 to 154.1] | 90 [40.2 to 103.6]
Statistical Analysis 1: Comparison: Arm I (Irinotecan, Cetuximab, Bevacizumab) vs Arm II (Irinotecan, Cetuximab, Placebo); Cetuximab comparison; Test type: Superiority; p = 0.4283, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Arm I (Irinotecan, Cetuximab, Bevacizumab) vs Arm II (Irinotecan, Cetuximab, Placebo); Irinotecan comparison; Test type: Superiority; p = 0.5262, Wilcoxon (Mann-Whitney)

11. Other Pre Specified Outcome: Change in Genotype Concentrations of Prespecified Gene Mutations in Circulating Cell-free Deoxyribonucleic Acid (DNA) (cfDNA)
Description: The mean and median change in mutation concentration for each prespecified gene, and provide the corresponding 95% confidence intervals will be estimated. Cox proportional hazards models will be applied to explore the predictive value of pretreatment mutation status for cetuximab sensitivity and resistance, using PFS and OS as the outcome variables.
Time Frame: Baseline up to 2 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Dynamic Change in Mutation Concentration While the Patient is Receiving Cetuximab Treatment
Description: Scatter plots and box plots will be used to illustrate such change.
Time Frame: Baseline up to 2 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 30 days from last dose of study treatment; Up to 51 months
Arm/Group | Arm I (Irinotecan, Cetuximab, Bevacizumab) | Arm II (Irinotecan, Cetuximab, Placebo)
All-Cause Mortality (participants affected / at risk) | 10/19 | 17/17
Serious Adverse Events (participants affected / at risk) | 5/19 | 5/17
Other Adverse Events (participants affected / at risk) | 19/19 | 17/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Irinotecan, Cetuximab, Bevacizumab) (N=19) | Arm II (Irinotecan, Cetuximab, Placebo) (N=17)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Fever (General disorders) | 0 (0) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Irinotecan, Cetuximab, Bevacizumab) (N=19) | Arm II (Irinotecan, Cetuximab, Placebo) (N=17)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 15 (164) | 12 (48)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 9 (62) | 7 (23)
Platelet count decreased (Investigations) | 5 (51) | 5 (18)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 15 (173) | 12 (61)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (14) | 0 (0)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (5)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (6)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 17 (213) | 15 (92)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14 (186) | 15 (96)
Hypertension (Vascular disorders) | 17 (193) | 13 (112)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-24): https://cdn.clinicaltrials.gov/large-docs/58/NCT02292758/Prot_SAP_000.pdf